CLINICAL TRIAL: NCT00392405
Title: Prevention of Contrast Induced Nephropathy With Sodium Bicarbonate
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Norton Community Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: A1
Record Dates: First submitted 2006-10-25; First posted 2006-10-26 (Estimated); Last update posted 2006-10-26 (Estimated); Status verified 2006-10

CONDITIONS: Contrast Induced Nephropathy
Keywords: Contrast Induced Nephropathy

INTERVENTIONS:
Drug: 3 amps of sodium bicarbonate mixed in one liter of D5W

SUMMARY:
This will be a randomized controlled trial closely following the original protocol in the previous study published in JAMA 2004 by Merten et al. Patients will be randomly assigned to one of two treatment groups. Treatment group A will receive 1cc/kg/hour of 0.9% normal saline at least 2 hours prior to study beginning and will be continued during and for 6 hours post contrast. Treatment group B will receive 3cc/kg of sodium bicarbonate solution for one hour prior to procedure then drip rate will be decreased to 1cc/kg/hour during and for 6 hours post procedure. The sodium bicarbonate solution will be made by adding 3 amps of bicarbonate to 1L of D5W. Patients in both treatment arms weighing >110kg the initial fluid bolus and drip will be limited to those patients weighing 110kg. In both treatment arms, diuretics will be held before and after contrast administration on the day of the study. BMP will be checked the day of, 24 and 48 hours post contrast administration. The greatest change in all readings will be used for treatment comparisons. Contrast induced nephropathy will be defined as a change in serum creatinine of more than 25% from baseline and/or 0.5mg/dL. Urinary pH will also be measured on first spontaneous void following bolus. Vital signs including blood pressure and oxygen saturation will be documented every 4 hours to monitor patients closely for signs and symptoms of volume overload

DETAILED DESCRIPTION:
Inclusion Criteria:

* Stage III Chronic Kidney Disease (GFR 30-60ml/min per 1.73m2 calculated by using MDRD equation)
* Inpatients at Norton Community Hospital scheduled to undergo diagnostic CT Scan using contrast between the hours of 7am and 6pm
* 18+ years of age

Exclusion Criteria

* Current clinical diagnosis of exacerbated congestive heart failure
* Creatinine >8 mg/dL
* Change in serum Cre of at least 0.5mg/dL during previous 24hours
* Pre-existing dialysis patient
* Multiple myeloma
* Uncontrolled hypertension (definition: treated SBP >160mmHg or DBP >100mmHg
* Exposure to contrast 48 hours prior to study
* Allergy to contrast dye
* Pregnancy
* Patient has received pressor agents, fendolapam, mannitol, or mucomyst at time of study
* Acute myocardial infarction

Subjects: Consecutive samples of all CPSC inpatients who meet the above inclusion criteria

Allocation Assignment: Patients who meet inclusion criteria and agree to participate in the study will pick a concealed number out of an open envelope. That number (between 1- 656) will correlate with a number on a sealed opaque envelope. Inside the opaque envelope will be a chart sticker. The chart sticker will have the words either normal saline or sodium bicarbonate. The envelope will not be opened until all patient information (ie. Patient ID sticker) is placed on the original chosen envelope. Then the chart sticker will be removed and placed on the chart

Protocol Outline:

This will be a randomized controlled trial closely following the original protocol in the previous study. Patients will be randomly assigned to one of two treatment groups. Treatment group A will receive 1cc/kg/hour of 0.9% normal saline at least 2 hours prior to study beginning and will be continued during and for 6 hours post contrast. Treatment group B will receive 3cc/kg of sodium bicarbonate solution for one hour prior to procedure then drip rate will be decreased to 1cc/kg/hour during and for 6 hours post procedure. The sodium bicarbonate solution will be made by adding 3 amps of bicarbonate to 1L of D5W. Patients in both treatment arms weighing >110kg the initial fluid bolus and drip will be limited to those patients weighing 110kg. In both treatment arms, diuretics will be held before and after contrast administration on the day of the study. BMP will be checked the day of, 24 and 48 hours post contrast administration. The greatest change in all readings will be used for treatment comparisons. Contrast induced nephropathy will be defined as a change in serum creatinine of more than 25% from baseline and/or 0.5mg/dL. Urinary pH will also be measured on first spontaneous void following bolus. Vital signs including blood pressure and oxygen saturation will be documented every 4 hours to monitor patients closely for signs and symptoms of volume overload

ELIGIBILITY:
Inclusion Criteria:

* Stage III Chronic Kidney Disease (GFR 30-60ml/min per 1.73m2 calculated by using MDRD equation)
* Inpatients at Norton Community Hospital scheduled to undergo diagnostic CT Scan using contrast between the hours of 7am and 6pm
* 18+ years of age

Exclusion Criteria:

* Exclusion Criteria
* Current clinical diagnosis of exacerbated congestive heart failure
* Creatinine >8 mg/dL
* Change in serum Cre of at least 0.5mg/dL during previous 24hours
* Pre-existing dialysis patient
* Multiple myeloma
* Uncontrolled hypertension (definition: treated SBP >160mmHg or DBP >100mmHg
* Exposure to contrast 48 hours prior to study
* Allergy to contrast dye
* Pregnancy
* Patient has received pressor agents, fendolapam, mannitol, or mucomyst at time of study
* Acute myocardial infarction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 656
Dates: Start 2006-11

PRIMARY OUTCOMES:
Development of contrast-induced nephropathy, defined as an increase in serum creatinine of 25% or more within 2 day after administration of contrast

SECONDARY OUTCOMES:
change in mean arterial pressure after initial bolus, mmHg
urine pH after initial bolus
contrast volume
change in serum bicarbonate
change in serum potassium
change in serum glucose
change in serum creatinine
change in estimated glomerular filtration rate
incidence of contrast induced nephropathy

CONTACTS AND LOCATIONS:
Overall Officials: Donna S Sanders, DO, Principal Investigator — Norton Community Hospital; Mathew Cusano, MD, Study Director — Norton Community Hospital
Locations (1):
- Norton Community Hospital, Norton, Virginia, United States

REFERENCES:
- [Background] Merten GJ, Burgess WP, Gray LV, Holleman JH, Roush TS, Kowalchuk GJ, Bersin RM, Van Moore A, Simonton CA 3rd, Rittase RA, Norton HJ, Kennedy TP. Prevention of contrast-induced nephropathy with sodium bicarbonate: a randomized controlled trial. JAMA. 2004 May 19;291(19):2328-34. doi: 10.1001/jama.291.19.2328. PMID 15150204
- [Background] Barrett BJ, Parfrey PS. Clinical practice. Preventing nephropathy induced by contrast medium. N Engl J Med. 2006 Jan 26;354(4):379-86. doi: 10.1056/NEJMcp050801. No abstract available. PMID 16436769